CLINICAL TRIAL: NCT06784089
Title: Relationship Between Fracture Type and Preoperative Nutritional Status with Postoperative Pain and Prognosis in Geriatric Hip Surgery
Brief Title: Relationship Between Fracture Type and Preoperative Nutritional Status with Postoperative Pain
Status: Recruiting | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ramazan Baldemir, specialist, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: 2024-BÇEK/193
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Nutrition; Postoperative Pain; Hip Fracture; Geriatric
Keywords: nutritional status; hip surgery.; geriatric patients; postoperative pain; postoperative prognosis
MeSH Terms: conditions — Pain, Postoperative; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Geriatric patients with hip fracture: Patients who are over the age of 65 and who will undergo surgery due to hip fracture and who agree to participate in this observational study and sign the informed consent form will be prospectively recorded using the patient follow-up forms we have prepared.
  Interventions: Other: Geriatric Nutrition Risk Index; Other: visual analog scale

INTERVENTIONS:
Other: Geriatric Nutrition Risk Index — GNRI will be calculated from the formula [1.489 X albumin (g/L)] + [41.7 (weight/ideal weight)]. If the patient's weight is more than their ideal weight, the weight/ideal weight ratio will be accepted as 1. The ideal weight will be calculated for men with the formula [(Height-100) -(Height-150/4)], for women with the formula [(Height-100) -(Height-150/2.5)]. According to the results, patients will be determined as no risk (GNRI > 98), low risk (92-98), severe/moderate risk (GNRI < 92).
  Other Names: GNRI
Other: visual analog scale — During the VAS evaluation, the patient will be asked to indicate the location of the pain on a 100 cm long scale where 0: no pain, 100: maximum pain, and the value shown by the patient will be recorded.
  Other Names: VAS

SUMMARY:
The geriatric patient group is a population that should be considered differently than other age groups due to physiological characteristics that change with age. When literature data is examined, it is seen that patients over the age of 65 are evaluated differently in studies. The rapid aging of the general population causes more elderly patients to need surgery. However, malnutrition is a common comorbidity in surgical patients . In addition, chronic diseases, multiple drug addiction, low nutritional intake, decreased appetite and psychological conditions seen in geriatric patients are risk factors for the development of nutritional deficiencies . Therefore, it is important to specifically consider geriatric patients, who frequently have these risk factors, in terms of malnutrition and to evaluate the nutritional status of these patients before surgery. It is estimated that the prevalence of malnutrition in hospitalized geriatric patients varies between 30% and 60%, depending on the population studied and the assessment tools applied . Despite these high malnutrition rates, this issue has not received sufficient clinical attention. Furthermore, malnutrition is highly associated with the prognosis of elderly perioperative patients, which may lead to poor clinical outcomes, increased morbidity and mortality, complication rates, decreased quality of life, prolonged hospital stay, and increased hospital and healthcare costs. A number of different screening tools are currently available to assess nutritional status in the elderly. However, there is currently no gold standard. The Nutrition Risk Score 2002 (NRS2002) is a nutritional screening tool for adult inpatients, launched in 2002 by the European Society of Clinical Nutrition and Metabolism (ESPEN). The Mini Nutritional Assessment - Short Form (MNA-SF), recommended by the European Union, and the Geriatric Nutrition Risk Index (GNRI), which has recently been evaluated as a new screening tool, has been validated for the diagnosis of malnutrition and the prediction of clinical outcomes, and is based on objective measurements that do not require patient cooperation, and whose validity has been demonstrated in other studies for the prediction of short- and long-term outcomes. In addition, the Prognostic Nutrition Index (PNI) is an indicator used to assess the nutritional status of surgical patients, estimate the risk of surgery, and make prognostic judgments. Although it has been stated that all four nutritional screening tools mentioned above can be used as prognostic indicators in geriatric surgical patients, the relationship between these screening tools and postoperative pain, complications, and hospital stay in geriatric patients undergoing orthopedic hip surgery has not yet been evaluated.

Hip fracture is a painful event that is frequently seen in older adults. Hip fractures are generally classified as femoral head fracture, femoral neck fracture, intertrochanteric fracture, and subtrochanteric fracture. Hip fracture is treated with proximal femoral nailing, partial hip replacement, and total hip replacement surgeries. Studies have reported that patients experience very high rates of moderate to severe pain following hip fracture surgery. This situation shows that the approach to pain management in hip surgery is still inadequate and that investigators need different perspectives on postoperative pain in these patients. It is known that hip fracture is associated with serious morbidity, mortality, and disability in the elderly. Inadequate pain management in these patients is associated with low motivation and has a high impact on functional recovery. Therefore, adequate pain management is important in patients with hip fractures to prevent mental and physical complications and to ensure appropriate compliance with rehabilitation. It is known that pain is affected by many factors such as biophysiological, biochemical, demographic, psychosocial, behavioral and moral variables and age. It is known that unmanaged postoperative pain will significantly affect cardiopulmonary and thromboembolic complications, morbidity and mortality, hospital discharge, quality of life and daily activities. In this context, determining the factors that predict acute pain will allow earlier intervention. Thus, short- and long-term morbidity, medication use, hospital stay and, accordingly, healthcare expenses will be reduced.This study aimed to evaluate the relationship between preoperative hip fracture type, surgery type, nutritional status and postoperative pain and prognosis (complications and hospital stay) in geriatric patients who will undergo hip surgery due to hip fracture. Secondly, it was aimed to determine which of the above-mentioned nutritional risk screening tools would be more appropriate in these patients and which nutritional risk screening tool could predict postoperative pain and prognosis in patients who will undergo hip surgery.

DETAILED DESCRIPTION:
Purpose/Hypothesis:

H0: There is no relationship between fracture type and preoperative nutritional status and postoperative pain and prognosis in geriatric hip surgery.

H1: There is a relationship between fracture type and preoperative nutritional status and postoperative pain and prognosis in geriatric hip surgery.

Material-Method:

This study will be conducted in accordance with the Declaration of Helsinki and will be conducted at the SBÜ Ankara Atatürk Sanatoryum Education and Research Hospital after receiving approval from the relevant units and ethics committee. The study was designed as a single-center prospective observational study.

Patients who are over the age of 65 and who will undergo surgery due to hip fracture and who agree to participate in this observational study and sign the informed consent form will be prospectively recorded using the patient follow-up forms investigators have prepared.

The standard anesthesia and analgesia protocol that investigators routinely apply to patients will be applied throughout the surgery. If the patient has pain after the surgery, the patient will not wait and the necessary analgesic treatment will be given to the patient. The patients' preoperative routine blood tests, age, height, body weight, BMI, gender, diagnoses, American Society of Anesthesiologists (ASA) physical status score, Charlson Comorbidity Index (CCI), fracture type (femoral head fracture, femoral neck fracture, intertrochanteric fracture, subtrochanteric fracture), surgery performed, duration of surgery, complications developed during the procedure or during postoperative follow-ups until discharge, Visual Analog Scale (VAS) at the first, second, fourth, eighth, sixteenth and twenty-fourth hours postoperatively will be recorded. During the VAS evaluation, the patient will be asked to show the location of their pain when evaluated as 0: no pain, 100: maximum pain on a 100 cm scale, and the value shown by the patient will be recorded.

During this process, additional analgesia treatment applied, if any, side effects such as headache, nausea-vomiting, hypotension, bradycardia, itching, sweating, respiratory depression due to analgesia treatment, and patient satisfaction will be recorded.

The malnutrition risk of the patients will be determined and the preoperative Nutritional Risk Score-2002 (NRS-2002), Albumin level, Prognostic Nutritional Index (PNI), GNRI, MNA-SF, Charlson Comorbidity Index (CCI) and the length of hospital stay of the patients will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hip surgery
* Patients with informed consent
* Patients over the age of 65
* Patients undergoing surgery with spinal anesthesia
* Patients evaluated in the ASA (American Society of Anesthesiologist) 1-2-3 category
* Those with a body mass index (BMI) between 18-35

Exclusion Criteria:

* Patients with ASA 4 and above
* Patients under the age of 65
* Those with a BMI below 18 and above 35,
* Patients with systemic inflammatory diseases,
* Patients using continuous anti-inflammatory/analgesic drugs,
* Patients with chronic pain before surgery,
* Those with pathological fractures,
* Multiple traumas
* Those with end-stage disease (malignancy),
* Severe renal failure, gastrointestinal ulceration or severe asthma that prevents the use of standard analgesia protocol
* Patients who have previously had hip surgery on the same side
* Patients who want to have surgery with general anesthesia
* Patients who need general anesthesia in addition to spinal anesthesia
* Those with a history of Pulmonary Thromboembolism

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who are over the age of 65 and who will undergo surgery due to hip fracture
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Relationship between preoperative nutritional status with postoperative pain | 24 hours
  The primary outcome variable of the study was to evaluate the correlation between preoperative nutritional status with postoperative pain, in geriatric patients undergoing hip surgery due to hip fracture.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Atatürk Sanatorium Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No